CLINICAL TRIAL: NCT02769663
Title: Cognitive Complaints in Obstructive Sleep Apnea
Status: Completed | Type: Observational
Sponsor: VieCuri Medical Centre (Other)
Collaborators: Tilburg University (Other); Reinier de Graaf Groep (Other)
Responsible Party: Principal Investigator, Tim Vaessen, klinisch neuropsycholoog, VieCuri Medical Centre
Other Study IDs: ABR 37795
Record Dates: First submitted 2016-05-09; First posted 2016-05-11 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Cognition Disorders; Sleep Apnea Syndromes, Obstructive
MeSH Terms: conditions — Cognition Disorders; Sleep Apnea Syndromes | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- OSA: Patients with newly diagnosed obstructive sleep apnea and no medical comorbidity affecting cognition.
  Interventions: Behavioral: questionnaires and neuropsychological assessments
- healthy controls: Participants with no sleep disorder or other medical comorbidity affecting cognition.
  Interventions: Behavioral: questionnaires and neuropsychological assessments

INTERVENTIONS:
Behavioral: questionnaires and neuropsychological assessments

SUMMARY:
The study assesses cognitive complaints in newly diagnosed patients with obstructive sleep apnea with no medical-comorbity affecting cognition. Cognitive complaints will be compared to healthy controls matched on age, sex and educational level. Factors related to cognitive complaints will also be assessed, including anxiety and depressive symptoms, complaints of fatigue and sleepiness, quality of life, psychological coping strategies and objective measures of cognition. Patients starting treatment for sleep apnea (continuous positive airway pressure or mandibular repositioning device) will be reassessed on all measures after 6 months of treatment to study the impact of treatment as usual on cognitive complaints and its related factors.

ELIGIBILITY:
Inclusion Criteria:

* native Dutch speaker
* estimated verbal-IQ of ≥80

Exclusion Criteria:

* other sleep disorder than obstructive sleep apnea
* substance or alcohol abuse (e.g. no more than three units of alcohol per day for males and no more than two units of alcohol per day for females
* diagnosis of a psychiatric disorder
* use of medication effecting cognition
* neurological disease, diabetes mellitus, hypo- or hyperthyroidism or lung disease (as checked by verbal report and medical records)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients newly diagnosed with obstructive sleep apnea according to the clinical guidelines of the adult OSA taskforce of the American Academy of Sleep Medicine (apnea/hypopnea-index (AHI) of ≥15 or AHI of ≥5 with significant daytime symptoms)
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2012-06-01; Primary Completion 2018-08-16 (Actual); Study Completion 2019-02-18 (Actual)

PRIMARY OUTCOMES:
Cognitive Failure Questionnaire (CFQ) | Assessed at inclusion of study and, if treatment is started, after 6 months of treatment.
  Questionnaire assessing cognitive complaints
Behavior Rating Inventory of Executive Function Adult version (BRIEF-A) | Assessed at inclusion of study and, if treatment is started, after 6 months of treatment.
  Questionnaire assessing cognitive complaints

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Assessed at inclusion of study and, if treatment is started, after 6 months of treatment.
  questionnaire assessing anxiety and depressive symptoms
Fatigue Assessment Scale (FAS) | Assessed at inclusion of study and, if treatment is started, after 6 months of treatment.
  questionnaire assessing fatigue
Epworth Sleepiness Scale (ESS) | Assessed at inclusion of study and, if treatment is started, after 6 months of treatment.
  questionnaire assessing sleepiness
Pittsburgh Sleep Quality Index (PSQI) | Assessed at inclusion of study and, if treatment is started, after 6 months of treatment.
  questionnaire screening for sleep disorders and assessing sleep quality
Sleep diary | Assessed at inclusion of study and, if treatment is started, after 6 months of treatment.
  subjective measure for sleep quality
World Health Organisation Quality of Life Questionnaire BREF (WHOQOL-bref) | Assessed at inclusion of study and, if treatment is started, after 6 months of treatment.
  questionnaire measuring quality of life
Utrechtse Coping Lijst (UCL) | Assessed at inclusion of study and, if treatment is started, after 6 months of treatment.
  questionnaire measuring psychological coping strategies
Dutch reading tests for adults (NLV) | Assessed at inclusion of study.
  cognitive test for verbal intelligence
Central Nervous System Vital Signs Symbol Digit Coding (CNS-VS-SDC) | Assessed at inclusion of study and, if treatment is started, after 6 months of treatment.
  cognitive test for attention
Central Nervous System Vital Signs Continuous Performance Test (CNS-VS-CPT) | Assessed at inclusion of study and, if treatment is started, after 6 months of treatment.
  cognitive test for attention
Central Nervous System Vital Signs Stroop Test (CNS-VS-ST) | Assessed at inclusion of study and, if treatment is started, after 6 months of treatment.
  cognitive test for attention/executive function
Central Nervous System Vital Signs Shifting Attention Test (CNS-VS-SAT) | Assessed at inclusion of study and, if treatment is started, after 6 months of treatment.
  cognitive test for attention/executive function
Rey Auditory Verbal Learning Test (RAVLT) | Assessed at inclusion of study and, if treatment is started, after 6 months of treatment.
  cognitive test for memory
Wechsler Adult Intelligence Scale III - Digit Span (WAIS-III-DS) | Assessed at inclusion of study and, if treatment is started, after 6 months of treatment.
  cognitive test for attention/executive function
Trail Making Test (TMT) | Assessed at inclusion of study and, if treatment is started, after 6 months of treatment.
  cognitive test for attention/executive function
Semantic Fluency | Assessed at inclusion of study and, if treatment is started, after 6 months of treatment.
  cognitive test for executive function

CONTACTS AND LOCATIONS:
Overall Officials: Margriet Sitskoorn, PhD, Study Director — Tilburg University
Locations (2):
- Netherlands (2):
  - VieCuri Medisch Centrum, Venlo, Limburg
  - Reinier de Graaf Gasthuis, Delft, South Holland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vaessen TJA, Mark RE, Overeem S, Sitskoorn MM. Cognitive complaints in obstructive sleep Apnea: The overlooked role of coping styles. Sleep Med. 2025 Oct;134:106695. doi: 10.1016/j.sleep.2025.106695. Epub 2025 Jul 17. PMID 40706402